CLINICAL TRIAL: NCT06730984
Title: Endoscopy-Assisted Tracheal Intubation Versus Conventional Tracheal Intubation for Endoscopic Submucosal Dissection (ESD): a Prospective Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-139A-02
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Tracheal Intubation; Endoscopic Submucosal Dissection; Endoscopy-Assisted; Video Laryngoscope

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopy-Assisted Tracheal Intubation (Experimental): Tracheal Intubation Under Endoscopic Guidance
  Interventions: Other: Endoscopy-Assisted Tracheal Intubation
- Traditional Tracheal Intubation (Active Comparator): Tracheal Intubation Under Video Laryngoscopy
  Interventions: Other: Traditional Tracheal Intubation

INTERVENTIONS:
Other: Endoscopy-Assisted Tracheal Intubation — Tracheal Intubation Under Endoscopic Guidance
  Arms: Endoscopy-Assisted Tracheal Intubation
Other: Traditional Tracheal Intubation — Tracheal Intubation Under Video Laryngoscopy
  Arms: Traditional Tracheal Intubation

SUMMARY:
This study plans to enroll 148 patients undergoing upper gastrointestinal endoscopic submucosal dissection (ESD). Patients will be randomly divided into a control group (conventional tracheal intubation) and an experimental group (endoscopy-assisted tracheal intubation). Patients meeting the inclusion criteria and not falling under the exclusion criteria will be invited to participate in the study. Upon providing voluntary consent, the research physician will arrange for the patient's inclusion in the study. After signing the informed consent form, the research physician will collect the patient's basic information, medical history, and other details, followed by timing the preoperative preparation period and evaluating postoperative discomfort

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endoscopic submucosal dissection (ESD) at Ningbo University Affiliated First Hospital from December 2024 to December 2026.
* Aged between 18 and 75 years.
* Patients who voluntarily agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Individuals under 18 years of age.
* Patinents unwilling or unable to provide informed consent.
* Patients with severe chronic cardiac or pulmonary disease, or those who have required hospitalization for coronary or cerebrovascular events or radiotherapy within the past 3 months.
* Patients with severe abdominal symptoms such as severe pain, bloating, or nausea.
* Patients with inadequate preoperative preparation.
* Individuals requiring lifelong anticoagulant therapy, those with severe bleeding disorders, or those who have recently taken anticoagulant or antiplatelet medications.
* Pregnant or breastfeeding individuals.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2026-12-08 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
preoperative preparation time | 10 mins
  the time from Initiate Anesthesia Induction to Insert the Therapeutic Endoscope into the Oral Cavity

SECONDARY OUTCOMES:
The time to view the vocal cords (TVVC) | 1 min
  the time from inserting the tracheal tube into mouth to the operator view the the entire vocal cords
The time to advance the tracheal tube into trachea (TATT) | 1 min
  the time from viewing the entire vocal cords to insert the tracheal tube into trachea successfully

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No